CLINICAL TRIAL: NCT04070625
Title: Evaluation of the Effectiveness of a Communication Book in Pragmatic Communication in Vascular Aphasics During the First Year Post-Stroke
Brief Title: Communication Book in Pragmatic Communication in Vascular Aphasics
Acronym: APHACOM
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2008/10
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Aphasia; Communication
MeSH Terms: conditions — Aphasia; Communication | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Communication book group: Speech therapy with communication book
  Interventions: Other: Communication book group
- Control group: Simple speech therapy
  Interventions: Other: Control group

INTERVENTIONS:
Other: Communication book group — Communication book
  Groups: Communication book group
Other: Control group — Simple speech therapy
  Groups: Control group

SUMMARY:
This study aims to evaluate, in communication tasks, the pragmatic effectiveness of the communication book in the general conditions of use and its maintenance in the implementation of the compensatory strategies of communication in severe aphasias.

DETAILED DESCRIPTION:
Data from the literature have demonstrated the effectiveness of speech therapy in aphasic vascular. In the face of sequelae, particularly in the most serious aphasia, a palliative approach aims to increase the functional effectiveness of communication in everyday life. The communication book has been developed in this perspective, addressing aphasics whose language communication skills are greatly reduced. Early use in this trial is warranted by implantation prior to the onset of potentially deleterious compensatory mechanisms seen in the late-stage aphasic sequelae.

This study aims to evaluate, in communication tasks, the pragmatic effectiveness of the communication book in the general conditions of use and its maintenance in the implementation of the compensatory strategies of communication in severe aphasias.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent after information. Information is also given to the person of trust when it exists.
* aphasic subjects admitted to hospital or seen in consultation following a 1st ischemic or hemorrhagic symptomatic vascular accident constituted
* during the first year of onset of aphasia
* adults over 18 years old
* French
* phasic disorder of severe severity expression (overall severity score between 0 and 2 at the diagnostic battery for the assessment of aphasia scale)
* residual ability to understand clinical assessments and informed consent; information about the objectives and the procedure of the research will also be given to the patient's designated confidant
* motor capacity for comfortable sitting and transfers with help
* affiliation to health insurance
* no deficits in visual perceptual tests (researched using the visual decision of objects and Montreal protocol for the evaluation of visual gnosis), which allows the use of the communication book,

Exclusion Criteria:

* refusal or impossibility of consent
* disturbance of vigilance
* insane state
* psychiatric history requiring hospitalization in a specialized environment
* perceptual disturbance, visual agnosia not allowing the use of the image support
* pregnancy or breastfeeding
* administration after the occurrence of stroke of a product for which an effect on the recovery of aphasia has been reported: piracetam, bromocriptine, donepezil, dextroamphetamine (if treatment with these products has been performed, inclusion is possible after a weaning period of 15 days)
* simultaneous inclusion in another therapeutic protocol of language disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the six participating neurological rehabilitation centers, each of which has significant recruitment of aphasic subjects and has a specialized team in the management of language disorders.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2009-02-17 (Actual); Primary Completion 2012-02-10 (Actual); Study Completion 2012-02-10 (Actual)

PRIMARY OUTCOMES:
Number of successful tasks in the communication book | At Day 45 after stroke
  Communication book of Gonzales et al, with 6 tasks
Number of successful tasks in the communication book | At Day 90 after stroke
  Communication book of Gonzales et al, with 6 tasks

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alain JOSEPH, Pr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No